CLINICAL TRIAL: NCT05314790
Title: Management of Patients With Diagnosis of Hypothyroidism, as Hospitalized and as Outpatients, in Internal Medicine Units: Observational Study Before & After Educational Programme
Acronym: TIAMO
Status: Completed | Type: Observational
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.05.2015
Record Dates: First submitted 2022-01-20; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group (CG): Without intervening Educational Program
- training group (TG): Group who has received an Educational Program (EP). The implementation of an EP based on meetings within the Department, coordinated by an outside tutor (outreach visit model). The EP content was defined beforehand by a Scientific Board, on the basis of evidence-based guidelines (EBGs) and an up-to-date literature review, but also with a specific focus on any departures from standard clinical practice recommendations (CPRs) identified at each IM department in phase 1.
  Interventions: Other: intervening Educational Program

INTERVENTIONS:
Other: intervening Educational Program — The implementation of an EP is based on meetings within the Department, coordinated by an outside tutor (outreach visit model). The EP content was defined beforehand by a Scientific Board, on the basis of evidence-based guidelines (EBGs) and an up-to-date literature review, but also with a specific focus on any departures from standard clinical practice recommendations (CPRs) identified at each IM department in phase 1;
  Groups: training group (TG)

SUMMARY:
There is still limited knowledge regarding the clinical profile and appropriateness of treatment in patients with hypothyroidism hospitalized in Internal Medicine (IM) Departments in Italy. The aim of this study is to evaluate: 1) the characteristics of patients and possible deviations from national and international clinical practice recommendations (CPRs) in evidence-based guidelines (EBGs); 2) the improvement of patient management by means of a standardized educational programme (EP).

Methods: A nationwide multicentre study, comprising two replications of a retrospective survey (phases 1 and 3) with an intervening EP (phase 2) in half of the centres and no EP in the other half, was conducted. The EP was based on outreach visits. Centres were assigned to the two arms of the study, labelled the training group (TG) and control group (CG) respectively, by cluster randomization.

DETAILED DESCRIPTION:
Hypothyroidism (HT) is a common disorder that affects more than 4% of the general population. Since this percentage does increase with advancing age, it is reasonable to suppose that hypothyroidism is becoming a widespread disease condition. Furthermore hypothyroidism is correlated with significant cardiovascular morbidity and mortality.

Although the potential clinical impact of hypothyroidism, the clinical profile of patients affected by hypothyroidism and managed in the Internal Medicine setting it is not very well known so far. This study has the aim to take a real-life picture of Internal Medicine patients with diagnosis of hypothyroidism, in order to evaluate possible deviations between the current clinical practice and the evidence-based guidelines, and possibly improving the management by means of an educational program.

The FADOI-TIAMO study is designed as a replicate of two cross-sectional surveys (Phase 1 and 3) interspersed with an educational program (Phase 2) to be conducted in 11 out of the 22 participating Centres. The data collection in Phases 1 and 3 will be based on the review of medical records of the last 30 consecutive patients with known or de novo diagnosis of HT observed in each Centre (globally, 1200 patients).

ELIGIBILITY:
Inclusion Criteria:

* known diagnosis of hypothyroidism on the basis of medical history or laboratory results, as indicated in the clinical record of inpatients admitted to the IM department for any condition

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with known diagnosis of hypothyroidism on the basis of medical history or laboratory results,as hospitalized and as outpatients, in Internal Medicine Units
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
To evaluate any possible offset between treatment standards for hypothyroidism and the real-life management of patient | 4 months for each phase
  To evaluate, in the real-life management of the hypothyroidism therapy, possible deviations from national and international clinical practice recommendations (CPR) in evidence-based guidelines (EBGs). Four EBGs and 39 CPRs have provided the basis on which 22 treatment management indicators have been identified (e.g. Number of Patients on LT4 replacement therapy who are not taking oral solution or softgel formulations are on absorption-hindering medication and/or do not comply with timing in relation to meals / Number of patients on LT4 replacement therapy who do not comply with the prescribed timing before meals and/or are taking absorption-hindering medication; Number of patients on replacement therapy with TSH in the ATA target range/ Number of patients on replacement therapy with known TSH; Number of patients on replacement therapy, taking LT4 tablets at least 60' before breakfast or at least 3 h after dinner / Number of patients on replacement therapy with LT4 tablets)
Effects of an educational programme | 4 months for each phase
  To evaluate the improvement of some indicators (the same of outcome 1) in the management of patients with hypothyroidism by means of a standardized educational programme (e.g. Number of Patients on LT4 replacement therapy who are not taking oral solution or softgel formulations are on absorption-hindering medication and/or do not comply with timing in relation to meals / Number of patients on LT4 replacement therapy who do not comply with the prescribed timing before meals and/or are taking absorption-hindering medication; Number of patients on replacement therapy with TSH in the ATA target range/ Number of patients on replacement therapy with known TSH; Number of patients on replacement therapy, taking LT4 tablets at least 60' before breakfast or at least 3 h after dinner / Number of patients on replacement therapy with LT4 tablets)

SECONDARY OUTCOMES:
Clinical profile evaluation of hypothyroidism | 4 months for each phase
  Assessment of age, gender, weight, hormonal hypothyroidism status (TSH, FT3, FT4), comorbidity, treatment of hypothyroidism and other pharmacological therapies of patients with hypothyroidism

CONTACTS AND LOCATIONS:
Overall Officials: MAURO CAMPANINI, Study Director — FADOI FOUNDATION
Locations (20):
- Italy (20):
  - ULSS1 Belluno San Martino, Belluno
  - Ospedale Versilia, Camaiore
  - Ospedale di Canicattì, Canicattì
  - Ospedale di Castiglione del Lago, Medicina del Trasimeno, Castiglione del Lago
  - Garibaldi Nesima, Catania
  - Ospedale G.B. Morgagni - P.L. Pierantoni, Forlì
  - Ospedale G.P. Delogu, Ghilarza
  - Ospedale Gubbio-Gualdo Tadino, Gubbio
  - Ospedale "F. Veneziale", Isernia
  - ASL Latina, Latina
  - Ospedale S. Andrea, Massa Marittima
  - Ospedale S. Croce di Moncalieri - ASL TO5, Moncalieri
  - Ospedale Del Mare, Napoli
  - Ospedale Fatebenefratelli, Napoli
  - Ospedale Maggiore di Novara, Novara
  - Ospedale Civico di Partinico, Palermo
  - Ospedale "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - AOU di Sassari, Sassari
  - Ospedale San Paolo, Savona

REFERENCES:
- [Derived] Brancato D, Biondi B, Attardo TM, Fierro A, Nizzoli M, Vettor R, Monaco E, Romano R, Ariete V, Usai C, Zagarri E, Campanini M. Management of Hypothyroidism in Internal Medicine: Patient Profile and Effects of an Educational Programme in the Cluster-Randomized FADOI TIAMO Study. Front Endocrinol (Lausanne). 2022 Jun 13;13:839300. doi: 10.3389/fendo.2022.839300. eCollection 2022. PMID 35769080